CLINICAL TRIAL: NCT00309231
Title: Clinical Islet Transplantation Using the Edmonton Protocol
Status: Withdrawn | Type: Observational
Why Stopped: no funding
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Dr. William Wall, Lawson Health Research Institute
Other Study IDs: R-05-873; 11898
Record Dates: First submitted 2006-03-29; First posted 2006-03-31 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2010-06

CONDITIONS: Type 1 Diabetes
Keywords: diabetes mellitus; islet transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Islet Allotransplantation — Clinical islet transplantation using the Edmonton protocol, steroid free immunosuppression using sirolimus and tacrolimus and basilixumab induction therapy

SUMMARY:
The purpose of this study is to perform a series of islet transplants using the Edmonton protocol. Patients with Type I Diabetes and glycemic lability, severe hypoglycemia or hypoglycemic unawareness will undergo transplantation of purified pancreatic islets from cadaveric donors into the portal vein, followed by steroid-free immunosuppression as per the Edmonton protocol (IL-2 antibody induction, sirolimus, low dose tacrolimus-based immunosuppression). The goals of the transplant are to improve glycemic control, stabilize blood sugars and achieve insulin independence.

DETAILED DESCRIPTION:
The purpose of this study is to document the outcomes of islet transplant at our centre while replicating the Edmonton protocol. The Edmonton protocol, as described above, is currently the standard clinical protocol for conducting clinical islet transplantation in selected patients with type 1 diabetes. We propose to conduct a feasibility study to document the availability and frequency of donor organs, test the process of islet isolation, assess the implementation of procedures to transplant islets and administer immunosuppression, monitor the complications of immunosuppression and document the success and safety of the transplant procedure at our centre.

The outcomes we propose to document include: 1) the number of patients who achieve insulin independence one year after completing the Edmonton protocol 2) the A1c value one year after completing the Edmonton protocol 3) graft survival as measured by basal and stimulated C-peptide levels 4) islet equivalents isolated from each donor organ and islet equivalents per kg transplanted 5) complications of islet transplant and immunosuppressive therapy.

Eight patients who have had type 1 diabetes for more than 5 years will undergo islet allotransplantation using the Edmonton protocol. It is expected that most patients will require a minimum of two transplant procedures to receive enough islets to achieve insulin independence. Procedures will follow published guidelines.

Pancreata will be isolated from brain-dead donors according to published protocols, including the two-layer cold storage method. Islets will be cultured for up to 48 hours to facilitate timing of the islet infusion.

Islets will be infused into the portal vein. Post transplant immunosuppression will consist of the modified Edmonton protocol as outlined by Ryan et al including basiliximab induction therapy, sirolimus and tacrolimus maintenance therapy, aspirin and enoxaparin thromboprophylaxis, pneumocystis carinii prophylaxis with sulfamethoxazole/trimethoprim for 6 months and cytomegalovirus prophylaxis for 3 months if indicated. Insulin requirements will be monitored closely after transplant. Serum glucose, glycosylated haemoglobin, serum C-peptide, creatinine, and lipid concentrations will be monitored.

Patients will be seen in follow up every month initially and longer term every 3 to 6 months as required. Glucose control, immunosuppressive levels and adverse events will be monitored regularly. Patients will be monitored for complications of diabetes as per standard guidelines. Tests of beta cell function (mixed meal Ensure test for glucose and C-peptide) will be performed every 3 months initially and then every 6 months once stable.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* type 1 diabetes for at least 5 years
* at least 1 of the following: a) frequent, severe hypoglycaemia b) hypoglycemic unawareness* c) glycemic lability despite an optimal insulin regimen*, and failure of intensive insulin therapy as judged by independent endocrinologist

Exclusion Criteria:

* obesity (BMI >28
* insulin requirements > 0.7 U/kg/day
* history of cancer (except basal or squamous skin cancer)
* unstable, severe, or non-correctable cardiac disease
* previous organ transplant
* evidence of sensitization (PRA>20%)
* renal dysfunction (macroalbuminuria, renal dialysis)
* untreated proliferative retinopathy
* active infection, including hep C, hep B, HIV, TB
* current cigarette smoking (6 months abstinence required) or substance abuse
* indication for steroid medications (exception steroid inhalers, topical steroids)
* indication for anticoagulation (exception aspirin)
* pregnancy or desire for future pregnancy; breast-feeding
* major psychiatric illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes of at least 5 years duration, with either severe hypoglycemia with unawareness, or severe glycemic lability
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Study Completion 2008-01

PRIMARY OUTCOMES:
Efficacy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William Wall, MD, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre University Campus, London, Ontario, Canada

REFERENCES:
- [Background] Ryan EA, Paty BW, Senior PA, Bigam D, Alfadhli E, Kneteman NM, Lakey JR, Shapiro AM. Five-year follow-up after clinical islet transplantation. Diabetes. 2005 Jul;54(7):2060-9. doi: 10.2337/diabetes.54.7.2060. PMID 15983207
- [Background] Shapiro AM, Lakey JR, Ryan EA, Korbutt GS, Toth E, Warnock GL, Kneteman NM, Rajotte RV. Islet transplantation in seven patients with type 1 diabetes mellitus using a glucocorticoid-free immunosuppressive regimen. N Engl J Med. 2000 Jul 27;343(4):230-8. doi: 10.1056/NEJM200007273430401. PMID 10911004
- [Background] Tsujimura T, Kuroda Y, Avila JG, Kin T, Oberholzer J, Shapiro AM, Lakey JR. Influence of pancreas preservation on human islet isolation outcomes: impact of the two-layer method. Transplantation. 2004 Jul 15;78(1):96-100. doi: 10.1097/01.tp.0000133515.37892.d5. PMID 15257045
- [Background] Lakey JR, Burridge PW, Shapiro AM. Technical aspects of islet preparation and transplantation. Transpl Int. 2003 Sep;16(9):613-32. doi: 10.1007/s00147-003-0651-x. Epub 2003 Aug 19. PMID 12928769